CLINICAL TRIAL: NCT04969328
Title: ParTNer-STEPs: Parents in Transition - a Nurse-led Support and Transfer Education Program
Brief Title: Parents in Transition - a Nurse-led Support and Transfer Education Program
Acronym: ParTNer-STEPs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Bente Appel Esbensen, Professor, Senior Researcher, RN, MSciN, Ph.D, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ParTNer-STEPs
Record Dates: First submitted 2021-06-30; First posted 2021-07-20 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Chronic Illness
Keywords: Adolescent; Chronically ill; Parents; Transitional care; Patient transfer
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: The study has a RCT design and consist of a intervention- and a control group (1:1).
  The study is part of a complex intervention design consisting of four phases: development, pilot testing, evaluation and implementation. The RCT study is together with a qualitative process evaluation part of the evaluation phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ParTNer-STEPs (Active Comparator): Parents and adolescents will receive the ParTNER-STEPs program and standard care.
  Interventions: Other: ParTNer-STEPs
- Standard care (No Intervention): The adolescent and their parents will receive standard care

INTERVENTIONS:
Other: ParTNer-STEPs — The intervention is a transfer program (ParTNer-STEPs), offered to the parents 1½ - ½ year before their child´s transfer to adult care.
  ParTNer-STEPs consist of
  1. an informative website available for parents from recruitment until follow-up.
  2. online educational events for parents. The teaching events are offered twice a year as a web based seminar with short presentations on different topics. The seminars will not be available for parents after their child has transferred to adult care.
  3. transfer consultations across the paediatric and adult department. The transition consultations consist of:
     * a preparatory consultation (3-6 months before transfer) with the paediatric nurse.
     * a farewell consultation with the paediatric nurse (0-3 months before transfer).
     * a joint consultation (at transfer) where both the pediatrician and the adult physician will be present.
     * a welcoming consultation with the nurse from the adult care (0-3 months after transfer).
  Arms: ParTNer-STEPs

SUMMARY:
OBJECTIVE To improve chronically ill adolescents' transition to adult care by preparing and supporting the parents. The study aim is to improve parents' (of chronically ill adolescents, 16-18 years) transition readiness by offering them a brief transition program.

HYPOTHESIS Young peoples´ self-management skills are mainly developed at home, guided by their parents, rather than in consultations with health professionals.

The investigators hypothesize that a nurse-led transfer intervention focusing on parents' knowledge, skills and attitudes will:

1. improve the parents´ readiness for their child's transition to adult health care
2. support the parents' gradual handing over of treatment responsibility to the adolescent and, that an improvement in parental transition readiness will
3. strengthen the adolescent's self-management skills and increase his/her readiness for transition.

BACKGROUND Transfer from paediatric to adult care for chronically ill adolescents is associated with no-shows and low treatment adherence, as well as anxiety and concerns among parents. Studies show that support for parents results in better transition for both parties.

INTERVENTION

ParTNer-STEPs is a transfer program consisting of three initiatives:

1. a website with information about the adult department and legal changes as well as advice from other parents and young people
2. online teaching events (web based seminars) for parents
3. transfer consultations across the paediatric and adult department

METHOD The intervention will be evaluated in a randomized controlled trial (RCT) study over two years. The project will be carried out in four paediatric outpatient clinics at Rigshospitalet, Copenhagen University Hospital, Denmark: nephrology, hepatology, neurology and rheumatology. Based on a power calculation, the investigators aim to include parents of minimum 62 adolescents. Primary outcome: Parents' transition readiness (TR). Secondary outcomes: Adolescents' TR, self-management skills, and quality of life.

DETAILED DESCRIPTION:
STUDY DESIGN The study design is a randomized controlled trail (RCT) study in a period of 6 to 18 months before the adolescent is transferred to adult care (depends on when the participant is recruited before transfer) and three months after transfer.

RECRUTMENT Potential participants will be contacted by the paediatric nurses at the four outpatient clinics and briefly informed of the study. If the parents are interested in the project, the project coordinator will provide the parents with oral and written information of the study, including the fact that they can withdraw from the study at any time without consequences for their child's treatment. There will also be provided written information to their adolescent child and the adolescent will also get the opportunity to speak directly to the project coordinator, if they have any questions. Finally, after time to consider their participation in the project, a written consent will be obtained. Under the recruitment process the investigators will carefully consider the risk of coercion, autonomy, and confidentiality.

RANDOMIZATION Randomisation will be conducted after screening and written consent of parents. Randomisation will by conducted by computer-generated (REDCap) random numbers as a dyad (adolescent and parents) with a ratio of 1:1 (using algorithm to stratify by the four outpatient's clinic). The dyads will be randomised into two groups 1) receive the intervention (standard care plus ParTNer-STEPs until their child´s transfer to adult care) or 2) standard care (control group). Once the database has defined a dyad's allocation, no changes can be made. Those randomised to the intervention arm will then receive access to the intervention materials.

SAMPLE-SIZE No previous studies have focused on whether it´s possible to increase parents´ transition readiness score (TR) by offering them a transfer program. A previous cross-sectional study found that parents of chronically ill adolescents have an average TR score of 3.12 (SD 0.68). Based on our clinical experience, advice from the author of the primary outcome questionnaire, and a review of each item in the questionnaire (Medical self-management and transition readiness), the investigators assume that it will be possible to increase the parents' TR score in the intervention group with 0,5 points.

The investigators are planning an RCT study with a continuous response variable from an independent control- and intervention group with 1 control(s) per intervention subject. Based on a previous study the investigators assume the response within each group will be normally distributed with standard deviation 0.68. If the true difference in the intervention and control means is 0.50, the investigators will need to include parents of 31 individual adolescents in each group to be able to reject the null hypothesis that the population means of the intervention and control groups are equal with probability (power) 0.80. The Type I error probability associated with this test of this null hypothesis is 0.05. Thus, the investigators need to recruit a total of parents of at least 62 individual adolescents.

SETTING The intervention will be carried out at the nephrology, hepatology, neurology and rheumatology paediatric and adult outpatient clinics at Copenhagen University Hospital, Rigshospitalet, Denmark. The investigators have chosen these four specialties, because low treatment adherence and non-attendance in the patient group could result in permanent disabilities or critical consequences. In Denmark adolescents transfer to adult care when turning 18 years old regardless of the adolescent's maturity or transitional readiness. Each paediatric clinic has at least one youth ambassador (a nurse with special interest and training in adolescent medicine). The existing transitional care includes youth consultations using the split-visit model and assessment of adolescent transition readiness. The clinics currently have no programmes targeting parents.

ETHICS The project will adhere to the regulations established by the Ethical Guidelines for Nursing Research in the Nordic Countries, all relevant laws and regulations in Denmark, and to the Declaration of Helsinki II and is approved by the Danish Data Protection Agency, reference no. VD-2018-396.

The investigators have formally enquired the regional research ethics committee with a full clinical description of the project. They have reviewed the project and given us permission to perform the study (reference no. FSP 20031083).

According to Danish legislation studies such as register research projects, interview surveys and questionnaire surveys can be performed without formal ethical approval cf. section 1 and 2 in the committee law as no human biological material is included.

Before obtaining consent from the parents, the investigator will provide all participants with oral and written information of the study, including the fact that they can withdraw from the study at any time without consequences for their child's treatment. The investigators will carefully consider the risk of coercion, autonomy, and confidentiality.

DATACOLLECTION Data will be collected though questionnaires at baseline and every six months up to three months after the adolescent's transfer to adult care. Questionnaires will be sent out via email or by post based on participants´ wishes.

DATA MANGEMENT All data will be handled confidential and stored in the password protected software REDCap.

DATA ANALYSIS A detailed statistical analysis plan (SOP) will be developed when all participants have completed the final measurement (six months after the completed intervention) in collaboration with statisticians. The investigators plan to include t tests, Pearson's Chi-square test, regression analysis, intention to treat and linear models. Logistic regression analyses will be carried out to describe transition readiness and allocation of responsibility within the intervention group and compare it to the control group's score. Socio-demographic data and the parents' uncertainty-score will be considered as variables. The SOP will be confirmed among all project group members before the investigators will be looking into data.

MISSING DATA, DROP OUT AND LOST TO FOLLOW UP Loss to follow-up and missing data for various reasons is impossible to avoid in randomized trials. The investigators will apply the analysis framework in which missing data related to the intention-to-treat approach depend on making plausible assumptions about the missingness of the data and including all participants in subsequent sensitivity analyses.

1. Attempt to follow up all randomized parents, even if they withdraw from allocated treatment.
2. Perform a main analysis of all observed data that are valid under a plausible assumption about the missingness of the data (i.e., Model-based: data as observed; using linear mixed effects models, assuming that data are 'Missing at Random' [MAR]).
3. Perform sensitivity analyses to explore the effect of departures from the assumption made in the main (#2) analysis (i.e., a non-responder-imputation: using the value at baseline to replace missing data will correspond to a non-responder imputation; these models will potentially be informative even if data are 'Missing Not At Random' [MNAR]).
4. Account for all randomized parents, at least in the sensitivity analyses (covered by #2 and #3 above, plus the corresponding analyses based on the per protocol population).

The interpretation of the corresponding statistical measures of uncertainty of the treatment effect and treatment comparisons will involve consideration of the potential contribution of bias to the P-value, 95% confidence interval, and of the inference in general.

Our primary analysis population will be all parents with available data at baseline, statistically modelled using repeated-measures linear mixed effects models (see above). These models will be valid if data are 'MAR'.

Sensitivity: The investigators will analyze all variables, with missing data being handled by multiple imputation techniques. When the different sensitivity analyses agree, and the analyses on the sensitivity analyses and the main analysis lead to essentially the same conclusions, confidence in the trial results is increased.

ELIGIBILITY:
Inclusion Criteria:

Parents, stepparents or guardians of chronically ill adolescents, who

* are aged 16.5-17.5 years (can be recruited up to six months before transfer)
* have been diagnosed for minimum six months
* have regular check-ups at the Department of Paediatrics and Adolescent Medicine's nephrology, hepatological, neurological and rheumatological outpatient clinics at Rigshospitalet, Denmark.
* are transferred to an adult hospital department
* are mentally and cognitively able to take responsibility for their own treatment

Exclusion Criteria:

* Parents who do not read and speak Danish
* Parents of adolescents who will be transferred to their family doctor at the age of 18 year.

Ages: 198 Months to 210 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Transition readiness (TR) | Change from baseline TR at transfer (last consultation in paediatrics)
  TR measured by the questionnaire Medical self-management and transition readiness. The questionnaire is validated. The questionnaire consists of 21 identically structured Likert-scaled items assessing the adolescent's awareness of their health condition and ability to make decisions relevant to their health care needs. All items ask participants to respond on a five item Likert-scale (1=strongly disagree, 2=disagree, 3= neither disagree nor agree; 4=agree and 5= strongly agree). Answered by parents (primary) and adolescent (secondary outcome)

SECONDARY OUTCOMES:
Allocation of Responsibility (AoR) | Change from baseline AoR at transfer (last consultation in paediatrics)
  AoR measured by the questionnaire Allocation of Responsibility. The questionnaire is validated and consists of 13 items. Participants answer questions on self-report measures. Respondents can choose from one of four answers: 1) parent/guardian takes primary responsibility, 2) responsibility is shared between the parent/guardian and the adolescent, 3) adolescent takes primary responsibility or 4) Not Applicable or No One Does This. Answered by parents and adolescents.
Uncertainty | Change from baseline uncertainty score at transfer (last consultation in paediatrics)
  Uncertainty measured by the uncertainty-scale. The scale is validated and measures parental uncertainty during transfer of their child from paediatric to adult care on a linear analogue scale from 0 (not uncertain at all) to 100 (extremely uncertain). Answered by parents
Health-related quality of life (HRQoL) | Change from baseline HRQoL at transfer (last consultation in paediatrics)
  HRQoL measured by EQ-5D-5L. The questionnaire comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. Answered by adolescents
Experiences of transfer | Three months after transfer (follow-up)
  Experiences of transfer measured by a self-developed questionnaire with 11 items based on modifiable factors from the SMART transition theory. All items ask participants to respond on a five item Likert-scale (1=strongly disagree, 2=disagree, 3= partially agree; 4=agree and 5= strongly agree). The questionnaire has been content and face validated by parents . Answered by parents
Transfer satisfaction | Three months after transfer (follow-up)
  Transfer satisfaction measured by a single question: 'On a scale of 0-100, how satisfied have participants been with their child's transition to the adult care?' The scale is a linear analogue scale from 0 (very unsatisfied) to 100 (very satisfied). Answered by parents and adolescents.

CONTACTS AND LOCATIONS:
Overall Officials: Bente A Esbensen, Professor, Principal Investigator — Center of Rheumatology and Spine Disorders, Copenhagen University Hospital, Rigshospitalet, Denmark
Locations (1):
- Center of Adolescent Medicine, Department of Paediatrics and Adolescent Medicine, Copenhagen University Hospital, Rigshospitalet, Denmark., Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Full dataset to replicate the analysis will be available from the corresponding author on reasonable request until five years after completion of the study, according to Danish law.

REFERENCES:
- [Background] Bilhartz JL, Lopez MJ, Magee JC, Shieck VL, Eder SJ, Fredericks EM. Assessing allocation of responsibility for health management in pediatric liver transplant recipients. Pediatr Transplant. 2015 Aug;19(5):538-46. doi: 10.1111/petr.12466. Epub 2015 Mar 31. PMID 25824486
- [Background] Burstrom A, Acuna Mora M, Ojmyr-Joelsson M, Sparud-Lundin C, Rydberg A, Hanseus K, Frenckner B, Nisell M, Moons P, Bratt EL. Parental uncertainty about transferring their adolescent with congenital heart disease to adult care. J Adv Nurs. 2019 Feb;75(2):380-387. doi: 10.1111/jan.13852. Epub 2018 Oct 18. PMID 30209810
- [Background] Schwartz LA, Brumley LD, Tuchman LK, Barakat LP, Hobbie WL, Ginsberg JP, Daniel LC, Kazak AE, Bevans K, Deatrick JA. Stakeholder validation of a model of readiness for transition to adult care. JAMA Pediatr. 2013 Oct;167(10):939-46. doi: 10.1001/jamapediatrics.2013.2223. PMID 23959392
- [Background] Williams T, Sherman E, Mah JK, et al. (2011) Measurement of medical self-management and transition readiness among Canadian adolescents with special health care needs. International Journal of Child and Adolescent Health 3: 527-535.
- [Background] Schwartz LA, Tuchman LK, Hobbie WL, Ginsberg JP. A social-ecological model of readiness for transition to adult-oriented care for adolescents and young adults with chronic health conditions. Child Care Health Dev. 2011 Nov;37(6):883-95. doi: 10.1111/j.1365-2214.2011.01282.x. PMID 22007989
- [Derived] Thomsen EL, Boisen KA, Hanghoj S, Hansson H, Grabow Scheelhardt HV, Christensen ST, Esbensen BA. A comprehensive transfer program from pediatrics to adult care for parents of adolescents with chronic illness (ParTNerSTEPs): study protocol for a randomized controlled trial. Trials. 2022 Dec 20;23(1):1034. doi: 10.1186/s13063-022-06997-0. PMID 36539857
- [Derived] Thomsen EL, Esbensen BA, Hanghoj S, Hansson H, Boisen KA. Development of a complex intervention to support parents of adolescents with chronic illness transferring from pediatrics to adult care (ParTNerSTEPs). BMC Health Serv Res. 2022 Apr 12;22(1):485. doi: 10.1186/s12913-022-07888-5. PMID 35413976

DOCUMENTS (1):
  • Study Protocol (2021-07-09): https://cdn.clinicaltrials.gov/large-docs/28/NCT04969328/Prot_000.pdf